CLINICAL TRIAL: NCT01259284
Title: A Double Blinded, Randomized Study Comparing the Effectiveness of Fish Oil Supplements, Oral Statins, and Placebo in Reducing the Incidence of Atrial Fibrillation Following a Lung Resection in Patients With Lung Cancer
Brief Title: Fish Oil Versus Statins Versus Placebos in Reducing Atrial Fibrillation in Patients Undergoing Thoracic Surgery for Lung Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0591
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancers
Keywords: Breast cancer; Colorectal cancer; Genitourinary cancer; Head and neck cancers; Lung cancer; Melanoma; Sarcoma; Atorvastatin; Lipitor; Fish Oil supplement; Placebo
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Urogenital Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Melanoma; Sarcoma | interventions — Atorvastatin; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Atorvastatin (Experimental): 1 Atorvastatin capsule daily plus 3 Placebo capsules twice a day orally, 5 days pre-surgery.
  Interventions: Drug: Atorvastatin; Other: Placebo
- Fish Oil Supplement (Experimental): 3 Fish Oil capsules twice a day plus 1 Placebo capsule daily orally 5 days pre-surgery.
  Interventions: Dietary Supplement: Fish Oil Supplement; Other: Placebo
- Placebo (Placebo Comparator): 4 capsules orally every morning and 3 every evening for 5 days pre-surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 1 capsule by mouth every morning 5 days before surgery, and 9 days after surgery or until discharge.
  Other Names: Lipitor
  Arms: Atorvastatin
Dietary Supplement: Fish Oil Supplement — 3 capsules by mouth in the morning and evening 5 days before surgery, and 9 days after surgery or until discharge.
  Other Names: n-3 PUFA; Fish oil supplementation
  Arms: Fish Oil Supplement
Other: Placebo — Placebo group: 4 capsules by mouth every morning and 3 every evening for 5 days before surgery and 9 days after surgery or until discharge.
  Atorvastatin group: 3 capsules by mouth every morning and evening, 5 days before surgery and 9 days after surgery or until discharge.
  Fish Oil Supplement group: 1 capsule by mouth every morning 5 days before surgery and 9 days after surgery or until discharge.

SUMMARY:
The goal of this clinical research study is to learn if Lipitor (atorvastatin) or fish oil supplements can help to control side effects of the heart that are commonly seen after lung surgery (such as irregular heartbeat). Researchers also want to learn if one of these drugs is more effective than the other at controlling side effects.

DETAILED DESCRIPTION:
The Study Drugs:

Atorvastatin is designed to lower cholesterol by blocking its production in the liver. This may help to decrease the chances of having a heart attack or a stroke.

Fish oil supplements are designed to lower fat levels in the blood by blocking their production in the liver. This may help to decrease the chances of having a heart attack or a stroke.

Atorvastatin is FDA-approved and commercially available for lowering cholesterol or fat levels in the blood. Fish oil supplements are also commercially available.

Researchers want to compare the anti-inflammatory effects of Atorvastatin and fish oil supplements.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study "Part" based on when you join this study. Up to 132 participants will be enrolled in Part 1 of the study. Up to 120 participants will be enrolled in Part 2 of the study.

If you are enrolled in Part 1, you will be randomly assigned (as in a roll of dice) to 1 of 3 groups. You will be provided with enough unmarked capsules for fourteen days plus a test dose. You will take the test dose in the clinic in the presence of the research nurse. Beginning 5 days before lung surgery (Day -5), you will take 1 capsule in the morning, as well as 3 capsules 2 time each day (a total of 7 unmarked capsules each day) for 5 days. The capsules should be taken with a cup (8 ounces) of water and may be taken with or without food. You will be reminded by the research nurse to bring the remaining capsules from home prior to your admission for surgery.

* If you are in Group 1, the capsules you will take will be fish oil supplements and placebo. A placebo is a substance that looks like the study drug but has no active ingredients.
* If you are in Group 2, the capsules you will take will be atorvastatin and placebo.
* If you are in Group 3, the capsules you will take will be placebo only.

You will have an equal chance of being assigned to each group. Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

After Part 1 is complete, the groups will be compared to learn if any group was more effective than the others. If neither fish oil supplements nor atorvastatin is shown to be more effective than the placebo, the study will be stopped. If fish oil or atorvastatin is found to be more effective than the placebo, the study will continue to Part 2.

If you are enrolled in Part 2, you will be randomly assigned to 1 of 2 study groups. You will be provided with enough unmarked capsules for fourteen days plus a test dose. You will take the test dose in the clinic in the presence of the research nurse, and begin taking capsules 5 days before surgery (Day -5) for 5 days. If atorvastatin was found to be the more effective drug in Part 1, you will take 1 unmarked capsule in the morning each day. If fish oil was found to be the more effective drug in Part 1, you will take 3 capsules 2 times each day (a total of 6 unmarked capsules each day). The capsules should be taken with a cup (8 ounces) of water and may be taken with or without food.

You will be reminded by the research nurse to bring the remaining capsules from home prior to admission for surgery.

* If you are in Group 1, the capsules you will take will be the drug that was found to be more effective in Part 1 (either fish oil supplements or atorvastatin).
* If you are in Group 2, the capsules you will take will be placebo only.

You will have an equal chance of being assigned to each group. Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Surgery:

After you have taken the study drug/placebo for 5 days, you will have standard of care lung surgery performed. You will be given a separate consent form to read and sign for the surgery.

On the day of surgery, any unused capsules will be collected and the days, times, and reasons why any doses were missed will be recorded. You will then continue taking the study drug/placebo for up to 9 days after surgery or until you are released from the hospital (whichever comes first). You will follow the same dosing schedule you followed before surgery.

Study Visits:

Each day while you are in the hospital, your vital signs will be measured and you will be checked for any allergic reaction you may have had to the study drug/placebo.

On Days 1 and 3, and on the last day that you take the study drug/placebo, blood (about 1 teaspoon) will be drawn to check your liver function.

About 4-6 weeks after surgery, you will have a follow-up visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any symptoms and/or side effects you may have had.
* Blood (about 1 teaspoon) will be drawn to check your liver function.

Length of Study:

You will take the study drug/placebo for 5 days before surgery, and for up to 9 days after surgery (up to a total of 14 days). Your participation in the study will be over after the follow-up visit. You will be taken off study early if you have intolerable side effects (such as allergic reaction or abnormal liver function tests).

This is an investigational study.

Up to 252 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients need to be in a normal sinus rhythm preoperatively.
2. Participants undergoing planned lobectomy and 60 years of age or older or participants undergoing planned pneumonectomy and 18 years of age or older.
3. Planned procedure is 5 days after the start of taking study drugs.
4. Signed written informed consent
5. Women of childbearing potential must have a negative pregnancy test (A woman of childbearing potential is a women who has not been naturally postmenopausal for at least 12 consecutive months or who has not undergone previous surgical sterilization)
6. Adequate liver function evidenced by; aspartate aminotransferase (AST or SGOT) </= 2.5 * Upper Limits of Normal (ULN), and alanine aminotransferase (ALT or SGPT) </= 2.5 * ULN

Exclusion Criteria:

1. Any history of supraventricular arrhythmia for which the patient is taking medications.
2. Current use of antiarrhythmic medications other than beta-receptor antagonists, calcium-channel antagonists, or digitalis.
3. Use of any supplemental n-3 fatty acids during the previous three months.
4. Use of any statin therapy during the previous three months.
5. Patients known to have a history of recent drug or alcohol abuse.
6. Known allergy to seafood
7. Current use of Gemfibrozil and Fenofibrate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Vaporciyan, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 06, 2011 to July 29, 2011. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: The study was terminated with only 2 participants enrolled. The inability to find participants was predominantly due to current or recent use of statins or fish oils.
Period: Overall Study
Arm/Group | Atorvastatin | Fish Oil Supplement | Placebo
Started | 2 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Study Termination | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Fish Oil Supplement | Placebo | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age Continuous [Mean (Full Range); unit: years] | 69 [68 to 70] |  |  | 69 [68 to 70]
Gender [Number; unit: participants]
  Female | 2 |  |  | 2
  Male | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidences of Atrial Fibrillation During First 4 Days After Lung Resection
Description: New onset of sustained (15 min or >) or clinically significant (requiring intervention) atrial fibrillation (AF) during first 4 days post surgery as defined by on American College of Cardiology and American Heart Association Physician Consortium.
Time Frame: Baseline to 4 days post surgery
Population: Analysis was to be per protocol. There is no analysis due to an inadequate number of enrolled participants in study which resulted in early termination.
Arm/Group | Atorvastatin | Fish Oil Supplement | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 Months
Arm/Group | Atorvastatin | Fish Oil Supplement | Placebo
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=2) | Fish Oil Supplement (N=0) | Placebo (N=0)
decreased hemoglobin (Blood and lymphatic system disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=2) | Fish Oil Supplement (N=0) | Placebo (N=0)
Pain in extremity (General disorders) | 1 | 0 | 0
hypotension (Blood and lymphatic system disorders) | 1 | 0 | 0
atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 1 | 0 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
fatigue (General disorders) | 1 | 0 | 0
anorexia (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No